CLINICAL TRIAL: NCT00136721
Title: Parkin Mutations and Their Functional Consequences
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: RBM03-48; DGS2004/0511 (Registry Identifier: N°ref DGS)
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2025-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; phenotype-genotype correlations; mutations spectrum; candidate genes
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients and controls seen in outpatients clinic were sampled, after signing an informed consent.

GROUPS / COHORTS (2):
- Parkinson: A large cohort of 655 patients with early-onset Parkinsons's disease (PD), 589 with late-onset PD and 390 patients with autosomal dominant PD have been sampled, according to the age at onset and family history.
- Paired controls: Setting up a collection of controls matched with patients for age, gender and geographic origin at each center

SUMMARY:
Parkinson's disease (PD) is the most frequent neurodegenerative disease with a prevalence of 2% over 65 years and because of this high prevalence as the population ages, it is a major problem of public health.

An exhaustive repertory of not only parkin mutations in autosomal recessive forms of PD but also in other known genes such as DJ-1, PINK1 and LRRK2, is of major importance for both genetic counseling in families affected with PD and physiopathological approaches to this disease.

Through a French network for the study of Parkinson's disease genetics and extended collaborations with European, Mediterranean and other various countries, a total of 2934 subjects including 1683 patients and 1251 unaffected individuals has been collected since 2002. These samples consisted of 122 families with autosomal recessive PD, 285 cases of isolated early onset PD, 110 autosomal recessive and 129 autosomal dominant families with late onset PD, 201 isolated late onset PD cases and 250 matched controls.

DNAs from all subjects are now available, lymphocytes and lymphoblastoid cell lines have been stored for most patients from France and recently, fresh fibroblasts have been obtained for some individuals.

The genetic approach to autosomal recessive PD is focused on the identification of mutations in the parkin gene but also on the screening of DJ-1, PINK1 and LRRK2 genes.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with Parkinson's disease, with a family history or not,
* Minors presenting clinical signs of the disease,
* Controls (without signs of the disease, matched by sex and age with the patients, relatives for the familial cases)

Exclusion Criteria:

* Persons refusing to sign the informed consent,
* Lack of clinical information

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Families with autosomal recessive PD, isolated early onset PD, autosomal recessive and autosomal dominant families with late onset PD, isolated late onset PD cases and matched controls.
Sampling Method: Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2005-02-08 (Actual); Primary Completion 2021-02-07 (Actual); Study Completion 2021-02-07 (Actual)

PRIMARY OUTCOMES:
Genetic analysis | Day 1
  On DNA extracted from a blood sample collected on EDTA and Lithium heparitane
Transcryptome analysis | Day 1
  On RNA extracted from a blood sample collected on PAX-Gene

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Brice, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris, University Paris 6
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Result] Lesage S, Magali P, Lohmann E, Lacomblez L, Teive H, Janin S, Cousin PY, Durr A, Brice A; French Parkinson Disease Genetics Study Group. Deletion of the parkin and PACRG gene promoter in early-onset parkinsonism. Hum Mutat. 2007 Jan;28(1):27-32. doi: 10.1002/humu.20436. PMID 17068781
- [Result] Lesage S, Janin S, Lohmann E, Leutenegger AL, Leclere L, Viallet F, Pollak P, Durif F, Thobois S, Layet V, Vidailhet M, Agid Y, Durr A, Brice A; French Parkinson's Disease Genetics Study Group; Bonnet AM, Borg M, Broussolle E, Damier P, Destee A, Martinez M, Penet C, Rasco O, Tison F, Tranchan C, Verin M. LRRK2 exon 41 mutations in sporadic Parkinson disease in Europeans. Arch Neurol. 2007 Mar;64(3):425-30. doi: 10.1001/archneur.64.3.425. PMID 17353388
- [Result] Foroud T, Pankratz N, Martinez M; PROGENI/GSPD-European Consortium. Chromosome 5 and Parkinson disease. Eur J Hum Genet. 2006 Oct;14(10):1106-10. doi: 10.1038/sj.ejhg.5201666. Epub 2006 May 31. PMID 16736031
- [Result] Rawal N, Periquet M, Lohmann E, Lucking CB, Teive HA, Ambrosio G, Raskin S, Lincoln S, Hattori N, Guimaraes J, Horstink MW, Dos Santos Bele W, Brousolle E, Destee A, Mizuno Y, Farrer M, Deleuze JF, De Michele G, Agid Y, Durr A, Brice A; French Parkinson's Disease Genetics Study Group; European Consortium on Genetic Susceptibility in Parkinson's Disease. New parkin mutations and atypical phenotypes in families with autosomal recessive parkinsonism. Neurology. 2003 Apr 22;60(8):1378-81. doi: 10.1212/01.wnl.0000056167.89221.be. PMID 12707451
- [Result] Periquet M, Latouche M, Lohmann E, Rawal N, De Michele G, Ricard S, Teive H, Fraix V, Vidailhet M, Nicholl D, Barone P, Wood NW, Raskin S, Deleuze JF, Agid Y, Durr A, Brice A; French Parkinson's Disease Genetics Study Group; European Consortium on Genetic Susceptibility in Parkinson's Disease. Parkin mutations are frequent in patients with isolated early-onset parkinsonism. Brain. 2003 Jun;126(Pt 6):1271-8. doi: 10.1093/brain/awg136. PMID 12764050
- [Result] Ibanez P, Lohmann E, Pollak P, Durif F, Tranchant C, Agid Y, Durr A, Brice A; French Parkinson's Disease Genetics Study Group. Absence of NR4A2 exon 1 mutations in 108 families with autosomal dominant Parkinson disease. Neurology. 2004 Jun 8;62(11):2133-4. doi: 10.1212/01.wnl.0000127496.23198.75. No abstract available. PMID 15184637
- [Result] Ibanez P, De Michele G, Bonifati V, Lohmann E, Thobois S, Pollak P, Agid Y, Heutink P, Durr A, Brice A; French Parkinson's Disease Genetics Study Group. Screening for DJ-1 mutations in early onset autosomal recessive parkinsonism. Neurology. 2003 Nov 25;61(10):1429-31. doi: 10.1212/01.wnl.0000094121.48373.fd. PMID 14638971
- [Result] Lucking CB, Chesneau V, Lohmann E, Verpillat P, Dulac C, Bonnet AM, Gasparini F, Agid Y, Durr A, Brice A. Coding polymorphisms in the parkin gene and susceptibility to Parkinson disease. Arch Neurol. 2003 Sep;60(9):1253-6. doi: 10.1001/archneur.60.9.1253. PMID 12975291
- [Result] Lohmann E, Periquet M, Bonifati V, Wood NW, De Michele G, Bonnet AM, Fraix V, Broussolle E, Horstink MW, Vidailhet M, Verpillat P, Gasser T, Nicholl D, Teive H, Raskin S, Rascol O, Destee A, Ruberg M, Gasparini F, Meco G, Agid Y, Durr A, Brice A; French Parkinson's Disease Genetics Study Group; European Consortium on Genetic Susceptibility in Parkinson's Disease. How much phenotypic variation can be attributed to parkin genotype? Ann Neurol. 2003 Aug;54(2):176-85. doi: 10.1002/ana.10613. PMID 12891670
- [Result] Lesage S, Durr A, Tazir M, Lohmann E, Leutenegger AL, Janin S, Pollak P, Brice A; French Parkinson's Disease Genetics Study Group. LRRK2 G2019S as a cause of Parkinson's disease in North African Arabs. N Engl J Med. 2006 Jan 26;354(4):422-3. doi: 10.1056/NEJMc055540. No abstract available. PMID 16436781
- [Result] Ibanez P, Lesage S, Lohmann E, Thobois S, De Michele G, Borg M, Agid Y, Durr A, Brice A; French Parkinson's Disease Genetics Study Group. Mutational analysis of the PINK1 gene in early-onset parkinsonism in Europe and North Africa. Brain. 2006 Mar;129(Pt 3):686-94. doi: 10.1093/brain/awl005. Epub 2006 Jan 9. PMID 16401616
- [Result] Leutenegger AL, Salih MA, Ibanez P, Mukhtar MM, Lesage S, Arabi A, Lohmann E, Durr A, Ahmed AE, Brice A. Juvenile-onset Parkinsonism as a result of the first mutation in the adenosine triphosphate orientation domain of PINK1. Arch Neurol. 2006 Sep;63(9):1257-61. doi: 10.1001/archneur.63.9.1257. PMID 16966503
- [Result] Brice A, Lohmann E, Ibanez P, Periquet M, Laine S, Debarges B, Lesage S, Dürr A. Phenotype/genotype correlations in Parkinson's disease. In: Relationships in Neurodegenerative Diseases, Cummings, Hardy, Poncet and Christen (Eds), Springer-Verlag Berlin Heidelberg Eds, 153-64, 2005.
- [Result] Lohmann E, Dürr A, Ruberg M, Brice A. Parkin. In: Parkinson's Disease: Genetic and Pathogenesis, Dawson Eds, in press, 2006.
- [Result] Brice A. [What can we learn from genes responsible for familial forms of Parkinson's disease?]. Bull Acad Natl Med. 2006 Feb;190(2):485-96; discussion 497-8. French. PMID 17001874
- [Result] Ishihara L, Warren L, Gibson R, Amouri R, Lesage S, Durr A, Tazir M, Wszolek ZK, Uitti RJ, Nichols WC, Griffith A, Hattori N, Leppert D, Watts R, Zabetian CP, Foroud TM, Farrer MJ, Brice A, Middleton L, Hentati F. Clinical features of Parkinson disease patients with homozygous leucine-rich repeat kinase 2 G2019S mutations. Arch Neurol. 2006 Sep;63(9):1250-4. doi: 10.1001/archneur.63.9.1250. PMID 16966502
- See also: Related Info — http://www.inserm.fr